CLINICAL TRIAL: NCT00143520
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled 26-week Dose-response Study of Rivoglitazone HCl (CS-011) With Active Comparator (Pioglitazone HCl) in Subjects With Type 2 Diabetes
Brief Title: Placebo and Active Controlled Study of Rivoglitazone in Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Medical monitor, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0011-203
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes
Keywords: Placebo and active control dose response study of rivoglitazone in type 2 diabetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rivoglitazone; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rivoglitazone
Drug: Pioglitazone
Drug: Placebo

SUMMARY:
This is a 6-month study to evaluate the effects of monotherapy with rivoglitazone, an insulin sensitizer, on glycemic control in newly identified type 2 diabetics or diabetics not adequately treated with other antidiabetic agents. The study tests rivoglitazone and uses a placebo and active treatment group for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes in male or female patients
* Between 18 and 75 years of age
* With a HbA1c greater than or equal to 7.5% and less than 10.5% at randomization

Exclusion Criteria:

* Type 1 diabetics or type 2 diabetics currently on insulin therapy
* Patients unwilling or unable to discontinue their anti-diabetic medication(s)
* History of ketoacidosis
* History of therapy with rosiglitazone, troglitazone, pioglitazone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2004-12; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c

SECONDARY OUTCOMES:
FPG, Lipids, hsCRP, Adiponectin

CONTACTS AND LOCATIONS:
Locations (74):
- United States (74):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Huntsville, Alabama
  - Muscle Shoals, Alabama
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Sherwood, Arkansas
  - Los Angeles, California
  - Moreno Valley, California
  - Sacramento, California
  - San Diego, California
  - San Mateo, California
  - Santa Monica, California
  - Torrance, California
  - Vista, California
  - West Hills, California
  - Newark, Delaware
  - Clearwater, Florida
  - Cocoa Beach, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Palm Harbor, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Warner Robins, Georgia
  - Chicago, Illinois
  - Gurnee, Illinois
  - Evansville, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Detroit, Michigan
  - Livonia, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Bozeman, Montana
  - Butte, Montana
  - Great Falls, Montana
  - Voorhees Township, New Jersey
  - Rochester, New York
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Marion, Ohio
  - Clinton, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Carrollton, Texas
  - Conroe, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Sugar Land, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Lakewood, Washington
  - Olympia, Washington
  - Renton, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Truitt KE, Goldberg RB, Rosenstock J, Chou HS, Merante D, Triscari J, Wang AC. A 26-week, placebo- and pioglitazone-controlled, dose-ranging study of rivoglitazone, a novel thiazolidinedione for the treatment of type 2 diabetes. Curr Med Res Opin. 2010 Jun;26(6):1321-31. doi: 10.1185/03007991003715079. PMID 20370378